CLINICAL TRIAL: NCT05443165
Title: The Effect of the Decision Support System Developed for Symptom Self-Management in Non-Hodgkin Lymphoma Patients on Symptom Management, Quality of Life, and Unplanned Hospital Admissions
Brief Title: The Effect of Decision Support System on Symptom Self-Management in Non-Hodgkin Lymphoma Patients
Acronym: LympSCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Merve Gözde SEZGİN, Principal Investigator, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 3890
Record Dates: First submitted 2022-06-28; First posted 2022-07-05 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Decision Support System; Non-Hodgkin Lymphoma
Keywords: Nursing; Decision Support System; Non-Hodgkin Lymphoma; Randomized Controlled Trial; Symptom Self-Management; Quality of Life
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Intervention Model Description: NHL patients meeting the sampling criteria will be assigned to the intervention and control groups by block randomization (1:1). NHL patients in the intervention group will be introduced to the decision support system regarding symptom self-management in face-to-face interviews. The decision support system will be asked to use it for three months on the 3rd, 7th, and 10th days of the 3rd, 4th and 5th chemotherapy cycles. A short SMS message will be sent to the patients on the 3rd, 7th, and 10th days of the 3rd, 4th and 5th chemotherapy courses. Participants will be able to contact researchers via the 24/7 contact button or by phone.
  In the control group, SMS will be sent to the control group on the 3rd, 7th, and 10th days after each chemotherapy to remind them about the frequency and severity of symptoms during the three-month follow-up. The "Lymphoma Patient Guide" link on the Turkish Society of Hematology page for the symptom management system will be sent to the patients via SMS.
Who Masked: Participant
Masking Description: Participants will be divided into groups according to the randomization list created to assign each patient to a group. Two independent researchers will conduct the assignment of participants to the intervention and control groups and the evaluation of outcome measurement data. Researchers will not be blinded as they make the interventions. However, participants will be blinded because they do not know the study's hypotheses and which group they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Symptom self-management with an online decision support system (Experimental): Symptom frequency and severity level of NHL patients will be evaluated with an online web-based application. NHL patients, who will be applying symptom self-management with an online decision support system, will be expected to additionally manage their symptom self-management using with this system. Participants in the intervention group will be asked to evaluate the frequency and severity of symptoms through the online symptom evaluation system on the 3rd, 7th, and 10th days of the 3rd, 4th, and 5th chemotherapy courses, and to use the decision support system for symptom self-management according to symptom severity. During the follow-up period, a short SMS message will be sent to the patients on the 3rd, 7th, and 10th days of the 3rd, 4th, and 5th chemotherapy cycles. In the third month, after the follow-up phase of the study is completed, the patients in the intervention group who come to the hospital for follow-up or treatment will receive post-tests.
  Interventions: Behavioral: The effectiveness of the online decision support system developed for symptom self-management
- Symptom self-management with an education booklet (Active Comparator): Symptom frequency and severity level of NHL patients will be evaluated with an online web-based application. NHL patients, who will be treated with the symptom self-management with education booklet. Participants will be asked to evaluate the frequency and severity of symptoms through the online symptom evaluation system on the 3rd, 7th, and 10th days of the 3rd, 4th, and 5th chemotherapy courses for three months. They will be able to do symptom self-management within the scope of the patient education booklet sent to them via SMS. During the follow-up period, a short SMS message will be sent to the patients on the 3rd, 7th, and 10th days of the 3rd, 4th, and 5th chemotherapy cycles. In the third month, after the follow-up phase of the study is completed, the patients in the intervention group who come to the hospital for follow-up or treatment will receive post-tests.
  Interventions: Behavioral: Symptom self-management with an education booklet

INTERVENTIONS:
Behavioral: The effectiveness of the online decision support system developed for symptom self-management — The online decision support system will appear with mild, moderate, or high severity according to symptom severity. If the patient's symptom is of mild category severity, a green area will appear on the screen and patients will see information on self-management strategies in this area. If patient's symptom is of moderate category severity, a yellow area will appear on the screen and patients will see information on self-management strategies and symptom monitoring at home in this area. In moderate symptom severity, when a yellow area occurs, patients should be asked, "Is your fever above 38℃?" according to their needs. Information about the treatment steps to be followed will be given. If the patient's symptom is in a severe category, a red area will appear on the screen and the patients will be warned to apply to the healthcare institution within this area.
  Arms: Symptom self-management with an online decision support system
Behavioral: Symptom self-management with an education booklet — Symptom frequency and severity level of NHL patients will be evaluated with an online web-based application. NHL patients, who will be treated with the symptom self-management with education booklet. Participants will be asked to evaluate the frequency and severity of symptoms through the online symptom evaluation system on the 3rd, 7th, and 10th days of the 3rd, 4th, and 5th chemotherapy courses for three months. They will be able to do symptom self-management within the scope of the patient education booklet sent to them via SMS.
  Arms: Symptom self-management with an education booklet

SUMMARY:
This study aims to evaluate the effect of the decision support system developed for symptom self-management on symptom management, quality of life, and unplanned hospital admissions in Non-Hodgkin lymphoma (NHL) patients. Since NHL patients often experience disease and treatment-related side effects after discharge from the hospital, it would be beneficial to develop web-based decision support systems that can support symptom management at home. A mobile-compatible symptom self-management decision support system will be developed and tested with five patients, based on the needs of NHL patients, evidence-based guidelines, and expert opinions. A randomized controlled trial design with a single-blind and active control group will be applied. NHL patients will be pretested and randomized (intervention: 26, control: 26). The intervention group will use the decision support system developed for symptom self-management for three months. The researchers will share their phone numbers with the patients and be contacted via the 24/7 contact button or the phone. The effectiveness of the decision support system developed for symptom self-management is planned to be evaluated at the beginning and after 12 weeks.

DETAILED DESCRIPTION:
Non-Hodgkin lymphoma (NHL) accounts for approximately 41% of the entire hematological cancer population. Improving symptom self-management of patients in NHL treatment and care is among the important goals. Symptom self-management in NHL patients is considered an important factor in the early detection and control of symptoms. Although treatment and care have an important role in the concept of symptom self-management in NHL patients, it is reported that the symptom self-management levels of the patients are generally low. Since NHL patients often experience disease and treatment-related side effects after discharge from the hospital, it seems necessary to develop web-based decision support systems that can support symptom management at home. Decision support system applications developed for symptom self-management; help patients manage their symptoms, coordinate treatment plans, receive comprehensive care, update their knowledge and encourage continuous learning. The study aims to evaluate the effect of the decision support system developed for symptom self-management in NHL patients on symptom management, quality of life, and unplanned hospital admissions.

In the study, a web-based decision support system for symptom self-management in NHL patients will be developed. The website content and decision support system will be prepared in line with current literature, national and international websites, and guidelines, evaluated with expert opinions and readability index, and will be finalized by testing with preliminary application. The study was designed as a randomized study with a single-blind and active control group. This study will be carried out with an NHL patient who is followed up and treated in the Hematology Outpatient Clinic and Daytime Chemotherapy Unit and meets the inclusion criteria of the sample. It will be prepared in line with the Consolidated Standard of Reporting Trials - CONSORT 2018 guidelines.

In the study, the sample size was calculated based on 80% power and 5% confidence interval on the G*POWER software package. The study will be conducted with cancer patients (n=52), 26 in the intervention group and 26 in the control group. Patients with NHL diagnosis (Diffuse Large B-Cell Lymphoma and Follicular Lymphoma), over 18 years of age, who received at least two cycles of chemotherapy, had an ECOG performance score of 0-1-2, were treated with chemotherapy for the first time due to NHL diagnosis and had no verbal communication disorder. Literate patients, have internet access, and use the internet will be included.

As a randomization method, the "block randomization method" will be chosen so that the participants in the intervention and control groups have similar characteristics. An independent researcher who was not involved in the research will be assigned to the intervention and control groups with the mobile application program. Randomization will be done in a computer environment using the http://www.r-bloggers.com/example-2014-2-block-/randomization/ website and put in opaque envelopes. After obtaining informed consent from patients who meet the inclusion criteria, pre-tests will be performed by the researcher. After the pre-tests are applied, the participants will be assigned to the groups with opaque envelopes prepared by an independent researcher. Thus, assignment bias will be prevented in the randomization process. As the participants do not know the hypothesis of the research and in which group they are, it will be ensured that the participants are blinded. For the patients in the control group not to understand the application to the intervention group, the link of the website prepared for the intervention group, which contains only information on the evaluation of symptom frequency and severity, will be opened to the patients in the control group with a password. Algorithms in the decision support system intervention protocol developed for symptom self-management to be tested in the intervention group will not be included in the website shared with the control group. Blinding the patients will be ensured by having a website that will be applied to both the intervention and control groups. Since the attempt is made by the researcher, the researcher cannot be blinded.

The decision support system designed for symptom self-management will be evaluated by experts, researchers by calculating the readability formula, and patients with NHL who will be included in the preliminary application. Pre-application will be made with NHL patients who meet the inclusion criteria and consent to participate in the study. It is aimed to make a preliminary application to 10% (n=5) of the sample. Patients who were taken into pre-application will not be included in the study.

A website for symptom self-management strategies of NHL patients will be developed. On the website, patients will be asked to evaluate the frequency and severity of symptoms with a visual analog scale. The severity of symptoms was categorized as mild, moderate, or severe in line with evidence-based guidelines; In line with the algorithms created according to the severity of the symptoms, the patients in the intervention group will be provided to use the decision support systems developed for symptom self-management. It is planned that the patients in the intervention group will use the decision support system for the evaluation of symptom frequency and severity and symptom self-management on the 3rd, 7th, and 10th days of the 3rd, 4th, and 5th chemotherapy courses. In addition, a short SMS message will be sent to the patients on the 3rd, 7th, and 10th days of the 3rd, 4th, and 5th chemotherapy cycles to remind the user of the decision support system developed for self-management. Three repeated SMS will be sent to patients who do not use the decision support system, and if the system is still not used, patients will be contacted by phone. Patients in the control group will benefit from routine hospital services for three months, and only the link of the website developed for symptom self-management strategies of NHL patients to evaluate symptom frequency and severity with a visual analog scale will be shared with patients. On the 3rd, 7th, and 10th days of the chemotherapy course, they will be asked to evaluate their symptom experience and severity. To remind the patients in the control group to evaluate the frequency and severity of symptoms, a short SMS message will be sent to the patients on the 3rd, 7th, and 10th days of the 3rd, 4th, and 5th chemotherapy cycles. In addition, the link to the "Lymphoma Patient Guide" on the Turkish Society of Hematology page for the symptom management system will be sent to the control group via SMS.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Diagnosed with NHL (Diffuse Large B Cell Lymphoma and Follicular Lymphoma)
* Chemotherapy for the first time due to the diagnosis of NHL
* Have received at least two cycles of chemotherapy
* ECOG performance score of 0-1-2
* Had no verbal communication disorder
* Literate
* Having internet access at home, having a device such as a tablet, computer, or phone, and being able to use these tools

Exclusion Criteria:

* Having metastases
* Undergoing major surgery
* With terminal disease
* ECOG performance score of 3 and above

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Rotterdam Symptom Checklist | 12 weeks
  The Rotterdam Symptom Checklist developed by De Haes et al. (1996) is used to evaluate the distress caused by the symptoms experienced by cancer patients. It consists of two sub-dimensions, Psychological and Physical Symptom. Scale items are scored on a Likert type ranging from one to four. The scale consists of 27 items in total, with the Psychological Symptom sub-dimension 8 items and the Physical Symptom sub-dimension 19 items. The Psychological Symptom subscale is the lowest 8 points, the highest 32 points, and the Physical Symptom subscale is the lowest 19 points and the highest 76 points. As the score obtained from the scale increases, the distress experienced also increases.
Functional Assessment of Cancer Therapy [FACT-G (Version 4)] Quality of Life Scale | 12 weeks
  The Functional Assessment of Cancer Therapy [FACT-G (Version 4)] Scale was developed by the "Center on Outcomes, Research and Education Northwestern Healthcare" headquartered in Evanston / Illinois in the United States, and the FACT-G (Version 4) evaluates the quality of life of malignant patients. FACT-G (Version 4) scales have been translated into many different languages. The scale items contain sentences evaluating the last week. A 5-point Likert-type scale (0: not at all, 1: very little, 2: a little, 3: quite a lot, 4: a lot) is used for the answers in the scale, which consists of 27 items. The total score is between 0-108. With FACT-G (Version 4), four dimensions of quality of life are evaluated: physical condition, social and family status, emotional status, and activity status. A high total score indicates that they perform their daily activities more.
Unplanned Hospital Applications Follow-up Form | 12 weeks
  As a result of the use of the decision support system developed for self-management of the patients in the intervention group, unplanned hospital admissions are expected to decrease. For this purpose, an Unplanned Hospital Application Form was prepared by the researchers to evaluate unplanned hospital admissions. With this form, unplanned hospital or emergency service admissions in the last three months, unplanned hospitalization, unplanned outpatient admission due to chemotherapy-related problems, and unplanned need for a new drug will be evaluated in patients with NHL in the intervention group. Each application frequency will be evaluated and the groups will be compared in this respect.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz Üniversitesi, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No